CLINICAL TRIAL: NCT06645730
Title: A Metabolomics-based Study of Predictors and Associated Mechanisms of Metabolic Disease Remission After Metabolic Syndrome Surgery.
Brief Title: Metabolomics Predictors for Metabolic Disease Remission After Metabolic Syndrome Surgery.
Status: Active, not recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dong Peng, Principal Investigator, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: 2024-223-01
Record Dates: First submitted 2024-10-14; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; metabolomics; hypertention; diabetes; fatty liver
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus; Fatty Liver | interventions — Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Metabolic syndrome combined with hypertension: Metabolic syndrome patients diagnosed with hypertension.
  Interventions: Diagnostic Test: hypertension
- Metabolic syndrome combined with diabetes: Metabolic syndrome patients diagnosed with diabetes.
  Interventions: Diagnostic Test: diabetes
- Metabolic syndrome combined with fatty liver: Metabolic syndrome patients diagnosed with fatty liver.
  Interventions: Diagnostic Test: fatty liver

INTERVENTIONS:
Diagnostic Test: hypertension — diagnosed with hypertension
  Groups: Metabolic syndrome combined with hypertension
Diagnostic Test: diabetes — diagnosed with diabetes
  Groups: Metabolic syndrome combined with diabetes
Diagnostic Test: fatty liver — diagnosed with fatty liver on CT
  Groups: Metabolic syndrome combined with fatty liver

SUMMARY:
Metabolic syndrome is a combination of several metabolic abnormalities that coexist, including obesity, insulin resistance, hypertension and dyslipidaemia. These metabolic abnormalities not only increase the risk of cardiovascular disease, but are also closely associated with metabolic diseases such as type 2 diabetes, fatty liver disease, and many types of cancer. With the prevalence of metabolic syndrome and its complications increasing year by year, how to effectively prevent and treat metabolic syndrome has become a major challenge for global public health. In recent years, metabolomics, as a high-throughput analytical technique to study metabolites in organisms, has been gradually applied to the study of metabolic syndrome and related metabolic diseases. Metabolomics can comprehensively depict the metabolic state of an organism and its dynamic changes, which provides a new perspective for revealing the pathological mechanisms of metabolic syndrome and searching for potential biomarkers. Through in-depth analysis of metabolomics data, researchers are able to better understand the complex pathological process of metabolic syndrome and provide a scientific basis for the development of personalised treatment and intervention strategies. Surgical intervention is a common treatment for patients with metabolic syndrome combined with metabolic diseases. However, postoperative metabolic status and disease remission are affected by a variety of factors, and the relevant mechanisms have not been fully clarified. Metabolomics-based approaches can systematically analyse the changes in metabolites before and after surgery, explore the key factors affecting postoperative remission, and reveal their underlying mechanisms. These studies can not only optimise the surgical treatment plan, but also provide an important theoretical basis for postoperative management.

DETAILED DESCRIPTION:
This study will include patients with a diagnosis of metabolic syndrome combined with one or more metabolic disorders (e.g., type 2 diabetes mellitus, fatty liver disease, hypertension, etc.) who are determined to be on the verge of undergoing relevant surgical procedures. Patients will be categorised into patients with comorbid hypertension, patients with comorbid diabetes mellitus and patients with comorbid fatty liver disease according to their comorbid metabolic diseases. Basic preoperative information was collected, and blood and stool were collected for hormone testing and metabolomics measurements before surgery. Comparison of metabolic disease remission after surgery was performed to evaluate the efficacy. To analyse the effects of preoperative and postoperative metabolomics and hormonal changes on metabolic disease remission in patients with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years;
* diagnosis of metabolic syndrome and combination of one or more metabolic diseases (e.g., type 2 diabetes mellitus, fatty liver disease, hypertension, etc.);
* identification of impending related surgical treatment;
* willingness to participate in this study and sign an informed consent form;
* complete clinical data.

Exclusion Criteria:

* Patients suffering from other serious systemic diseases (e.g., severe heart disease, renal insufficiency, liver cirrhosis, etc.) or malignant tumours;
* patients with acute diseases such as acute infections, acute myocardial infarction, acute stroke, etc.;
* patients who are on medications that may significantly affect their metabolic status (e.g., hormonal drugs, potent immunosuppressants, etc.);
* patients who cannot ensure compliance or are unwilling to cooperate with the study requirements;
* patients with Serious psychological disease or cognitive dysfunction, unable to understand the content of the study or cooperate with the study operation;
* Incomplete clinical data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients diagnosed with metabolic syndrome and undergoing bariatric surgery at the study centre.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Metabolic disease remission | From date of surgery until the date of first documented postoperative complication, assessed up to 2 months after surgery.
  Metabolic disease remission was defined as any remission of hypertention, diabetes, or fatty liver measured 2 months after surgery. Hypertension remission was defined as arterial blood pressure less than 140/90 mmHg measured postoperatively in patients with preoperative comorbid hypertension. Diabetes remission was defined as fasting blood glucose less than 6 mmol/L measured postoperatively in patients with preoperative comorbid diabetes. Fatty liver remission was defined as liver function in the normal range measured by postoperative blood tests in patients with preoperative comorbid fatty liver.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No